CLINICAL TRIAL: NCT05315271
Title: Comparative Study Between Ketamine-Bupivacaine Versus Bupivacaine With Intravenous Ketamine Infusion In Supraclavicular Brachial Plexus Block During Upper Limb Surgeries
Brief Title: Supraclavicular Brachial Plexus Block During Upper Limb Surgeries
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Abdelah, Resident of Anesthesiology , Intensive care unit and Pain management., Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: soh-Med-21-10-07
Record Dates: First submitted 2022-03-08; First posted 2022-04-07 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-05

CONDITIONS: Brachial Plexus Block
Keywords: Bupivacaine; ketamine; Brachial Plexus Block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): All patients will be randomly allocated into two equal groups: each group will contain 30patients:
  Interventions: Drug: Bupivacaine-ketamine injection
- Group 2 (Active Comparator): All patients will be randomly allocated into two equal groups: each group will contain 30patients:
  Interventions: Drug: Bupivacaine injection with intravenous ketamine infusion

INTERVENTIONS:
Drug: Bupivacaine-ketamine injection — 20 ml volume bupivacaine only (0.5%concentration) (with maximum dose not exceeding 4mg/kg ) plus ketamine (1 mg/kg) with maximum dose 100mg ; the total volume is 30 ml with the infusion of 100 ml normal saline at a rate of 100ml/h.
  Arms: Group 1
Drug: Bupivacaine injection with intravenous ketamine infusion — 20 ml volume bupivacaine only (0.5%concentration) (with maximum dose not exceeding 4mg/kg ) plus 10 ml saline ; the total volume is 30 ml with the infusion of ketamine 0.15 mg/kg added to 100 ml normal saline and will be infused at a rate of 100 ml/h, which will be stopped 5 min before the end of surgery.
  Arms: Group 2

SUMMARY:
Comparative Study Between Ketamine-Bupivacaine Versus Bupivacaine With Intravenous Ketamine Infusion In Supraclavicular Brachial Plexus Block During Upper limb Surgeries The techniques of regional anesthesia have become very popular as they provide several advantages in comparison with general anesthesia and systemic analgesia.

They provide perfect pain control, decreased complications and reduced post-anesthesia care unit stay.

Regional anesthesia provides more patient safety and better outcomes, which leads to the fact that ultrasound-guided regional anesthesia became more popular.

Ultrasound provides clinicians with real-time images which are useful for better identification of the anatomical structures, safe needle placement and adequate local anesthetic spread.

Brachial plexus blocks are commonly achieved via an interscalene, supraclavicular, infraclavicular or axillary approach.

The supraclavicular level is an ideal site to achieve anesthesia of the entire upper extremity just distal to the shoulder as the plexus remains relatively tightly packed at this level, resulting in a rapid and high-quality block. For this reason, the supraclavicular block is often called the ''spinal of the arm'' Using the local anesthetics alone for supraclavicular brachial plexus block provide good operative conditions but have the disadvantage of shorter duration of postoperative analgesia. Various adjuvants such as opioids, dexmedetomidine, dexamethasone, midazolam, ketamine, etc., were added to local anesthetics in brachial plexus block to achieve quick and prolonged block.

Ketamine is a noncompetitive antagonist of the N-methyl-D aspartate receptor(NMDAR).

It is used as a premedication, and for sedation, induction and maintenance of general anesthesia.

Local anesthetic and analgesic properties have been reported for ketamine. Intravenous administration of low-dose ketamine decreases postoperative opioid use and improves analgesia.

Ketamine has been added to bupivacaine to prolong the duration of regional anesthesia and postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years.
* ASA physical status I-II, scheduled.
* Patients of either sex.
* Unilateral elective upper limb surgeries undergoing under ultrasound guided supraclavicular brachial plexus block.

Exclusion Criteria:

* Patient refusal.
* Patients with peripheral neuropathy of the upper limb.
* Infection at the injection site.
* Uncontrolled diabetes, epilepsy, obstructive pulmonary disease and neuromuscular disease.
* Altered mental status.
* Hypersensitivity to bupivacaine and ketamine.
* Patients with coagulopathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Comparison of the efficacy of adding ketamine to bupivacaine versus intravenous ketamine infusion with supraclavicular brachial plexus block in upper limb surgeries of sensory block | 24 hours
  -Sensory block will be assessed by pin prick test using a 3-point scale : Grade 0 = normal sensation. Grade 1 = loss of sensation of pin prick (analgesia). Grade 2 = loss of sensation of touch (anesthesia).
  * Onset of sensory block: the time interval between the end of local anesthetic administration and complete sensory block by min.
  * Duration of sensory block: the time interval between the complete sensory block and complete resolution of anesthesia.
  Intraoperative: sensory block level will be assessed by a pin prick at in the dermatomal areas corresponding to the median, radial, ulnar, and musculocutaneous nerves every 15 minutes at (15 min, 30 min, 45 min ,60 min, Etc.) till end of the operation.
  Postoperative: will be checked every 30minutes until regain of pinprick sensation at (1/2hr, 1hr, 1.5hr and2hr) then at (3hrs, 6hrs, 12hrs and 24hrs).

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Abdallah F, Brull R Facilitatory effects of perineural dexmedetomidine on neuraxial and peripheral nerve block: a systematic review and meta-analysis. Br J Anaesth 110(6):915-925,2013. 2. Hanumanthaiah D, Vaidiyanathan S, Garstka M, Szucs S, Iohom G Ultrasound guided supraclavicular block. Med Ultrason 15(3):224-229,2013. 3. Argiriadou KS, McEwen A, Matthew G: Ultrasound-Guided Supraclavicular Brachial Plexus Block https: //www.wfsahq.org/components/com_virtual_library/media/2ffc0a053d75e1cae94f9 3f57cddb8ff-atow-384-00-01.pdf,2018. 4. Swami SS, Keniya VM, Ladi SD, et al. Comparison of dexmedetomidine and clonidine (α2 agonist drugs) as an adjuvant to local anaesthesia in supraclavicular brachial plexus block: a randomised double-blind prospective study. Indian J Anaesth; 56:243-249,2012. 5. Kohli S, Kaur M, Sahoo S, et al. Brachial plexus block: comparison of two different doses of clonidine added to bupivacaine. J Anaesthesiol Clin Pharmacol; 29:491-495, 2013. 6. Reves JG, Glass PS, Lubarsky DA, et al. Intravenous anesthetic. In: Miller R, editor. Miller's anesthesia. 7th ed. Philadelphia: Churchill Livingstone; 724-726, 2010.